CLINICAL TRIAL: NCT05080764
Title: A Randomized, Double Blind, Vehicle-controlled, Multicenter Phase II Study to Evaluate the Safety and Efficacy of BF-200 ALA (Ameluz®) and BF-RhodoLED® in the Treatment of Moderate to Severe Acne Vulgaris in Adults With Photodynamic Therapy (PDT)
Brief Title: Study to Evaluate the Safety and Efficacy of BF-200 ALA (Ameluz®) and BF-RhodoLED® in the Treatment of Moderate to Severe Acne Vulgaris With Photodynamic Therapy in Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biofrontera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALA-ACV-CT014
Record Dates: First submitted 2021-09-09; First posted 2021-10-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acne Vulgaris
Keywords: ALA-PDT
MeSH Terms: conditions — Acne Vulgaris | interventions — 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- 1h incubation BF-200 ALA (Experimental): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid) red light photodynamic therapy (PDT) utilizing BF-RhodoLED® after 1h incubation.
  Interventions: Combination Product: 1h Incubation Photodynamic therapy (PDT) (ALA-PDT, Ameluz®-PDT)
- 3h incubation BF-200 ALA (Experimental): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid) red light photodynamic therapy (PDT) utilizing BF-RhodoLED® after 3h incubation.
  Interventions: Combination Product: 3h Incubation Photodynamic therapy (PDT) (ALA-PDT, Ameluz®-PDT)
- 1h incubation vehicle (Placebo Comparator): Topical application of vehicle to BF-200 ALA red light photodynamic therapy (PDT) utilizing BF-RhodoLED® after 1h incubation.
  Interventions: Combination Product: 1h Incubation Photodynamic therapy (PDT) (vehicle to BF-200 ALA containing no active ingredient)
- 3h incubation vehicle (Placebo Comparator): Topical application of vehicle to BF-200 ALA red light photodynamic therapy (PDT) utilizing BF-RhodoLED® after 3h incubation.
  Interventions: Combination Product: 3h Incubation Photodynamic therapy (PDT) (vehicle to BF-200 ALA containing no active ingredient)

INTERVENTIONS:
Combination Product: 1h Incubation Photodynamic therapy (PDT) (ALA-PDT, Ameluz®-PDT) — The treatment field (whole face excluding the periocular area) will be cleansed with gauze soaked with ethanol or isopropanol. Afterwards, approximately 1 tube of study medication will be applied as a thin layer. After drug application, subjects should stay inside for 1 hour. Post incubation, red light illumination with BF-RhodoLED® will be performed according to the lamps user manual until a total light energy of 37 J/cm2 was applied. To cover the whole face 2 illuminations will be required which can either be performed subsequentially or in parallel (with 2 lamps).
  Other Names:
  ALA-PDT, Ameluz®-PDT
  Arms: 1h incubation BF-200 ALA
Combination Product: 1h Incubation Photodynamic therapy (PDT) (vehicle to BF-200 ALA containing no active ingredient) — The treatment field (whole face excluding the periocular area) will be cleansed with gauze soaked with ethanol or isopropanol. Afterwards, approximately 1 tube of study medication will be applied as a thin layer. After drug application, subjects should stay inside for 1h. Post incubation, red light illumination with BF-RhodoLED® will be performed according to the lamps user manual until a total light energy of 37 J/cm2 was applied. To cover the whole face 2 illuminations will be required which can either be performed subsequentially or in parallel (with 2 lamps).
  Arms: 1h incubation vehicle
Combination Product: 3h Incubation Photodynamic therapy (PDT) (ALA-PDT, Ameluz®-PDT) — The treatment field (whole face excluding the periocular area) will be cleansed with gauze soaked with ethanol or isopropanol. Afterwards, approximately 1 tube of study medication will be applied as a thin layer. After drug application, subjects should stay inside for 3 hours. Post incubation, red light illumination with BF-RhodoLED® will be performed according to the lamps user manual until a total light energy of 37 J/cm2 was applied. To cover the whole face 2 illuminations will be required which can either be performed subsequentially or in parallel (with 2 lamps).
  Other Names:
  ALA-PDT, Ameluz®-PDT
  Arms: 3h incubation BF-200 ALA
Combination Product: 3h Incubation Photodynamic therapy (PDT) (vehicle to BF-200 ALA containing no active ingredient) — The treatment field (whole face excluding the periocular area) will be cleansed with gauze soaked with ethanol or isopropanol. Afterwards, approximately 1 tube of study medication will be applied as a thin layer. After drug application, subjects should stay inside for 3h. Post incubation, red light illumination with BF-RhodoLED® will be performed according to the lamps user manual until a total light energy of 37 J/cm2 was applied. To cover the whole face 2 illuminations will be required which can either be performed subsequentially or in parallel (with 2 lamps).
  Arms: 3h incubation vehicle

SUMMARY:
The aim of this study is to test the safety and efficacy of photodynamic therapy (PDT) for the medication Ameluz® performed with the PDT-lamp BF-RhodoLED® in comparison to the respective placebo treatment for moderate to severe Acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability of the subject to provide informed consent and to sign the Health Insurance Portability and Accountability Act (HIPAA) form. A study-specific informed consent and HIPAA form must be obtained in writing prior to starting any study procedures. Minors under 18 years of age must be accompanied by the parent(s) or legal guardian(s) at the time of consent signing. The parent(s) or legal guardian(s) must also provide informed consent/HIPAA for the subject.
2. Subjects with moderate to severe acne on the face (IGA ≥3).
3. Presence of ≥20 inflammatory and ≥20 non-inflammatory (open and closed comedones) Acne vulgaris lesions on the face (should be located within not more than 2 illumination areas) as assessed by investigator.
4. All sexes, ≥16 years of age.
5. Willingness and ability to comply with study procedures, particularly willingness to receive up to 3 PDTs within 8 to 10 weeks.
6. Subjects with good general health or with clinically stable medical conditions will be permitted to be included in the study.
7. Willingness to stop topical facial treatments other than medical cleansers (i.e. face washes etc.) at least 14 days prior to randomization visit (Visit 2, baseline) and discontinue medical cleansers in the face at least 1 week prior to randomization visit (Visit 2, baseline) and thereafter until the end of study (use of soap is allowed but the product used should not be changed during the study).
8. Females of reproductive potential must have a negative serum pregnancy test and must use an adequate and highly effective or two effective methods of contraception throughout the study. (If hormonal contraception is used, the same product and dose should be taken for at least 6 months before the first treatment and throughout the entire study.)

Exclusion Criteria:

1. Any known history of hypersensitivity to ALA, porphyrins or excipients of BF-200 ALA.
2. History of soy or peanut allergy.
3. Subjects with sunburn or other possible confounding skin conditions (e.g. wounds, irritations, bleeding or skin infections) within or in close proximity (< 5 cm distance) to treatment field. (Reassessment of subjects is allowed once if the sunburn or other confounding skin conditions is/are expected to resolve within the screening period.

   Reassessment can be done on the day of the actual treatment.)
4. Clinical diagnosis of atopic dermatitis and other cutaneous conditions (e.g. lupus erythematosus), Bowen's disease, BCC, eczema, psoriasis, acne conglobate, acne fulminans, or secondary acne (steroid-induced acne, perioral dermatitis, acne rosacea), squamous cell carcinoma, other malignant or benign tumors in the treatment field.
5. Clinically significant (CS) medical conditions making implementation of the protocol or interpretation of the study results difficult or impairing subject's safety such as:

   1. Presence of photodermatoses or porphyria
   2. Metastatic tumor or tumor with high probability of metastasis
   3. Infiltrating skin neoplasia (suspected or known)
   4. Unstable cardiovascular disease (New York Heart Association class III, IV)
   5. Unstable hematologic (including Myelodysplastic syndrome), hepatic, renal, neurologic, or endocrine condition
   6. Unstable collagen-vascular condition
   7. Unstable gastrointestinal condition
   8. Immunosuppressive condition
   9. Presence of clinically significant inherited or acquired coagulation defect
6. Beard or other facial hair that might interfere with the study assessments unless subject agrees to be clean-shaven throughout the entire study period. (Reassessment of subjects is allowed once if assessment of acne lesions is impaired by facial hair at screening. Reassessment can be performed on the day of the actual treatment).
7. Facial procedures such as dermabrasion, chemical or laser peels as well as exposure to UV radiation (other than sunlight) at least 4 weeks prior to randomization visit (Visit 2, baseline).
8. Presence of strong artificial pigmentation (e.g. tattoos) or any other abnormality that may impact lesion assessment or light penetration in the treatment field.
9. Suspicion of drug or alcohol abuse.
10. Any topical medication of the skin prior to screening as defined below:

    1. Topical treatment with ALA or ALA-esters (e.g. MAL) or an investigational drug in- and outside the treatment field within 8 weeks prior to screening.
    2. Topical treatment with immunosuppressive, cytostatic or cytotoxic drugs inside the treatment field within 8 weeks prior to screening.
    3. Start of a regular and continuous topical administration of medication with hypericin or other drugs with phototoxic or photoallergic potential inside the treatment field within 4 weeks prior to screening. Subjects may, however, be eligible if such medication was regularly applied for more than 4 weeks prior to screening visit without evidence of an actual phototoxic/photoallergic reaction or if such medication is only administered for a limited time (e.g. an antibiotic)
11. Any use of the below specified systemic treatments within the designated periods:

    1. Systemic acne therapy (oral antibiotics within 8 weeks or oral isotretinoin within 6 months or start with hormonal therapy for acne within 6 months prior to Visit 2).
    2. Use of cytotoxic or cytostatic drugs within 6 months, or immunosuppressive therapies or use of ALA or ALA-esters (e.g. MAL) within 12 weeks, investigational drugs or drugs known to have major organ toxicity within 8 weeks, interferon or glycocorticosteroids (oral or injectable) within 6 weeks prior to screening.
    3. Start of long-term intake of medication with hypericin or systemically acting drugs with phototoxic or photoallergic potential within 8 weeks prior to screening. Subjects may, however, be screened and randomized if such medication was taken in or was regularly applied for more than 8 weeks prior to screening visit without evidence of an actual phototoxic/photoallergic reaction or if such a drug is only used for a limited time (e.g. an antibiotic).
12. Breast feeding women.
13. Subject unlikely to comply with protocol, e.g. inability to return for visits, unlikely to complete the study, or inappropriate in the opinion of the investigator.
14. Prior randomization in the study.
15. A member of study site staff or sponsor staff directly involved in the conduct of the protocol or a close relative thereof.
16. Simultaneous participation in a further clinical study.
17. Four or more nodular acne lesions on the face.
18. Unwillingness or inability to limit sun exposure for 48 hours post PDT treatment.

Dosing Day exclusion criteria:

1. Febrile or infectious disease within 7 days prior to PDT visits.
2. Subjects with sunburn, wounds, irritations, bleeding or other confounding skin conditions within illumination areas at PDT visits.
3. Application of topical glycocorticosteroids in- and outside the treatment field within 7 days prior to PDT visits
4. Administration of (topical or systemic) medication with phototoxic/photoallergic potential for a limited time. After discontinuing the medication, a wash out period of the medications 5-fold half-life time should be applied prior to the next PDT.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Relative change in the number of inflammatory lesions (relative change from baseline) 8 weeks after the last PDT as assessed by investigator. | 8 weeks after the last PDT
  Outcome 1 is the relative change in the number of inflammatory lesions at the final visit with respect to baseline as assessed by the investigator.
Treatment success defined by a minimum improvement of the modified investigator global assessment (mIGA) score by at least 2 assessed 8 weeks after the last PDT and resulting in an mIGA score of 0 (clear) or 1 (almost clear). | 8 weeks after the last PDT
  Treatment success is defined as a minimum improvement of the mIGA score by at least 2 and resulting in an mIGA score of 0 (clear) or 1 (almost clear).

SECONDARY OUTCOMES:
Absolute and/or percentage change from baseline in the number of lesions as assessed by investigator. | 4 or 8 weeks after the last PDT
  In particular, the following will be assessed:
  1. Inflammatory lesions - 4 weeks after the last PDT
  2. Inflammatory lesions - 8 weeks after the last PDT
  3. Non-inflammatory lesions - 4 weeks after the last PDT
  4. Non-inflammatory lesions - 8 weeks after the last PDT
  5. Inflammatory & non-inflammatory lesions - 4 weeks after the last PDT
  6. Inflammatory & non-inflammatory lesions - 8 weeks after the last PDT
Absolute and percentage change from baseline in the number of lesions as assessed by investigator. | 4 or 8 weeks after the last PDT
  In particular, the following will be assessed:
  1. Inflammatory lesions - 4 weeks after PDT-1
  2. Non-inflammatory lesions - 4 weeks after PDT-1
  3. Inflammatory and non-inflammatory lesions - 4 weeks after PDT-1
  4. Inflammatory lesions - 4 weeks after PDT-2
  5. Non-inflammatory lesions - 4 weeks after PDT-2
  6. Inflammatory and non-inflammatory lesions - 4 weeks after PDT-2
  7. Inflammatory lesions - 4 weeks after PDT-3
  8. Non-inflammatory lesions - 4 weeks after PDT-3
  9. Inflammatory and non-inflammatory lesions - 4 weeks after PDT-3
  10. Inflammatory lesions - 8 weeks after PDT-3
  11. Non-inflammatory lesions - 8 weeks after PDT-3
  12. Inflammatory and non-inflammatory lesions - 8 weeks after PDT-3
Absolute and percentage change from baseline in the number of lesions as assessed by investigator, only for responders at Visit 3 / 4 weeks after PDT-1. | 4 or 8 weeks after PDT-1
  In particular, the following will be assessed:
  1. Inflammatory lesions - 4 weeks after PDT-1
  2. Inflammatory lesions - 8 weeks after PDT-1
  3. Non-Inflammatory lesions - 4 weeks after PDT-1
  4. Non-Inflammatory lesions - 8 weeks after PDT-1
  5. Inflammatory & non-inflammatory lesions - 4 weeks after PDT-1
  6. Inflammatory & non-inflammatory lesions - 8 weeks after PDT-1
Absolute and percentage change from baseline in the number of lesions as assessed by investigator, only for responders at Visit 4b / 4 weeks after PDT-2. | 4 or 8 weeks after PDT-2
  In particular, the following will be assessed:
  1. Inflammatory lesions - 4 weeks after PDT-2
  2. Inflammatory lesions - 8 weeks after PDT-2
  3. Non-Inflammatory lesions - 4 weeks after PDT-2
  4. Non-Inflammatory lesions - 8 weeks after PDT-2
  5. Inflammatory & non-inflammatory lesions - 4 weeks after PDT-2
  6. Inflammatory & non-inflammatory lesions - 8 weeks after PDT-2
Absolute and percentage change in the number of lesions as assessed by investigator, only for responders at Visit 5b / 4 weeks after PDT-3. | 4 or 8 weeks after PDT-3
  In particular, the following be assessed:
  1. Inflammatory lesions - 4 weeks after PDT-3
  2. Inflammatory lesions - 8 weeks after PDT-3
  3. Non-Inflammatory lesions - 4 weeks after PDT-3
  4. Non-Inflammatory lesions - 8 weeks after PDT-3
  5. Inflammatory & non-inflammatory lesions - 4 weeks after PDT-3
  6. Inflammatory & non-inflammatory lesions - 8 weeks after PDT-3
Change in the number of nodules & cysts | 8 weeks after the last PDT
  Absolute change and percentage change from baseline (Visit 2) as assessed by investigator.
Treatment success defined by a minimum improvement of the IGA by at least 2. | 8 weeks after the last PDT
  Treatment success is defined as a minimum improvement of the IGA score by at least 2 (from baseline (Visit 2) as assessed by investigator).
Improvement of the IGA. | 8 weeks after the last PDT
  As assessed by the investigator.
Improvement of the mIGA. | 8 weeks after the last PDT
  As assessed by the investigator.
Improvement of scar severity and overall esthetic appearance. | 8 weeks after last PDT
  As assessed by the investigator via a physical global scale for acne scars (PGA)
Satisfaction regarding esthetic outcome and treatment. | 8 weeks after the last PDT.
  As reported by the subject.

OTHER OUTCOMES:
Frequency and severity of adverse events (AEs), serious AEs (SAEs), AEs of special interest (AESI) and treatment-emerged adverse events (TEAEs). | from screening to study completion, over a duration of up to approximately 25 weeks
  TEAEs are defined as all AEs with onset or worsening after first treatment with IMP up to the last visit of the subject (approximately 8 weeks post last PDT).
Application site skin reactions assessed by the investigator. | from screening to study completion, over a duration of up to approximately 25 weeks
  Application site skin reaction categories: discharge, erosion, erythema, exfoliation, fissure, induration, oedema, scabbing, skin flaking, ulceration, vesicles, other; severity of AE: mild, moderate or severe
Application site discomfort reported by the subjects. | from screening to study completion, over a duration of up to approximately 25 weeks
  pplication site discomfort categories: burning, hyperaesthesia, pain, paraesthesia, pruritus, stinging, warmth, other; severity of AE: mild, moderate or severe
Pain during illumination reported by the subject. | from screening to study completion, over a duration of up to approximately 25 weeks
  Assessed by the subjects using an 11-point numeric rating scale, where a score of 0 means "no pain" and a score of 10 means "worst imaginable pain".
Changes in blood pressure | at all clinic visits conducted over a duration of approximately 25 weeks
  systolic & diastolic [mmHg]
Changes in heart rate | at all clinic visits conducted over a duration of approximately 25 weeks
  [bpm]
Investigation of clinical chemistry parameters | first and last visit conducted up to approximately 25 weeks apart
  Findings which differ from reference range and are considered to be clinically significant are to be reported.
Investigation of hematology parameters | first and last visit conducted up to approximately 25 weeks apart
  Findings which differ from reference range and are considered to be clinically significant are to be reported.
Investigation of urinalysis parameters | first and last visit conducted up to approximately 25 weeks apart
  Findings which differ from reference range and are considered to be clinically significant are to be reported.
Physical examination of head, neck, skin, lymph nodes, thorax including heart and lungs, abdomen, and musculoskeletal, peripheral vascular and nervous system status | first and last visit conducted up to approximately 25 weeks apart
  Abnormal findings, considered to be clinically significant, are to be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc.
Locations (9):
- United States (9):
  - First OC Dermatology, Fountain Valley, California
  - Cosmetic Laser Dermatology, San Diego, California
  - Dermatology Associates PA of the Palm Beaches, Delray Beach, Florida
  - ForCare Clinical Research, Tampa, Florida
  - DelRicht Research, Baton Rouge, Louisiana
  - Skin Search of Rochester, Inc, Rochester, New York
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - DermResearch PA, Austin, Texas
  - Austin Institute for Clinical Research Inc., Pflugerville, Texas